CLINICAL TRIAL: NCT01725412
Title: Prevention of Renal Complications of Diabetes With Thiamine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Gudrun Caspar-Bell, Endocrinologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio REB #12-59
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Thiamine Supplementation (Experimental)
  Interventions: Dietary Supplement: Thiamine 300mg PO once daily
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Thiamine 300mg PO once daily
  Arms: Thiamine Supplementation
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
Thiamine is a key component in the creation of physiologic anti-inflammatory mediators. Serum thiamine stores have been found to be deficient in diabetic patients. Thiamine deficiency may be a key pathological mechanism of inflammation that results in diabetic kidney and retinal injury. The investigators hypothesize that the repletion of a patient's thiamine by oral supplementation may result in reduced inflammation, and therefore reduced kidney injury.

DETAILED DESCRIPTION:
Thiamine (vitamin B1) is a water-soluble vitamin. It is absorbed from the gastrointestinal tract and taken up into tissues by transport proteins and converted to thiamine pyrophosphate (TPP) by thiamine pyrophosphokinase (TPPK). TPP is a co-factor of pyruvate dehydrogenase (PDH), α-ketoglutarate dehydrogenase and transketolase (TKT)-enzymes involved in the metabolism of glucose.

Various transport proteins are involved in the transport of thiamine monophosphate (TMP) and TPP across membranes. These include thiamine transported isoform-1 (THTR1) and thiamine transporter isoform-2 (THTR2), reduced folate carrier-1 (RFC-1), which transports TMP and TPP across cell plasma membranes and the mitochondrial TPP transporter (mTHTR). Thiamine and TMP/TPP transporters may have abnormal expression in diabetes. Increased THTR1 levels are found in red blood cells (RBCs) and mononuclear leucocytes of patients with diabetes compared to those of healthy subjects. RBC precursors and leucocytes appeared to up-regulate THTR1 expression in response to decreased thiamine availability. In the presence of hyperglycemia, renal tubular epithelial cells, by contrast, have decreased expression. In both experimental models of diabetes and in human diabetics increased clearance of thiamine has been demonstrated. This precedes the development of microalbuminuria. Patients with microalbuminuria and early decline in glomerular filtration rate had higher fractional excretion of thiamine compared to patients with stable renal function.

Thiamine supplementation in STZ- diabetic mice prevented the development of microalbuminuria, decreasing urinary albumin excretion (UAE) by approximately 80%. In addition thiamine supplementation prevented diuresis and glycosuria. Human studies are limited but in one placebo controlled study the thiamine group showed a significant decrease in microalbuminuria in diabetic patients on thiamine.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of Type II diabetes which has been present for at least 5 years,
* persistent microalbuminuria (30-299 mg/24 h),
* HbA1c ≤ 8%, and
* BMI 19-40 kg/m2.

Exclusion Criteria:

* significant comorbidities,
* "deficient renal function" known allergy or intolerance to thiamine,
* use of thiamine supplements,
* participation in an interventional study within 30 days,
* recipients of renal and/or pancreatic transplant and
* women who were pregnant or breast feeding.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Microabluminuria

SECONDARY OUTCOMES:
Serum Thiamine Level

OTHER OUTCOMES:
Urinary Thiamine Level
Inflammatory Markers
  E-selectin, Intercellular Adhesion Molecule 1, von Willebrand Factor, malondialdehyde, glutathione, homocysteine, isoprotein F21, advanced glycation endproducts, receptor for advanced glycation endproducts

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Gudrun Caspar-Bell, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada